CLINICAL TRIAL: NCT06454188
Title: A Randomized, Placebo-controlled, Multicenter, Study to Evaluate the Impact of Upadacitinib on Spondyloarthritis Outcomes in Patients With Active Psoriatic Arthritis (UP-SPOUT)
Brief Title: A Study to Evaluate the Impact of Upadacitinib on Spondyloarthritis Outcomes in Patients With Active Psoriatic Arthritis
Acronym: UP-SPOUT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: CARE ARTHRITIS LTD. (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B24-033
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Psoriatic Arthritis; Spondyloarthritis, Axial
MeSH Terms: conditions — Arthritis, Psoriatic; Axial Spondyloarthritis | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Upadacitinib (Experimental): Participants randomized to this arm will receive Upadacitinib 15 mg tablets, once per day, for 12 weeks.
  Interventions: Drug: Upadacitinib 15 MG [Rinvoq]
- Placebo (Placebo Comparator): Participants randomized to this arm will receive matching placebo tablets with no active ingredients, once per day, for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Upadacitinib 15 MG [Rinvoq] — 15mg tablet once per day.
  Other Names: Rinvoq
  Arms: Upadacitinib
Drug: Placebo — 15mg tablet once per day.
  Arms: Placebo

SUMMARY:
A Randomized, Placebo-controlled, Multicenter, Study to Evaluate the Impact of Upadacitinib on Spondyloarthritis Outcomes in Patients with Active Psoriatic Arthritis (UP-SPOUT)

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥18 of age at the screening visit.
2. Subject must be able to understand and willing to adhere to all protocol requirements and voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/institutional review board (IRB), prior to the initiation of any screening or study-specific procedures.
3. Diagnosis of PsA by their treating rheumatologist.
4. Classification of PsA according to the CASPAR criteria19: Inflammatory articular disease (joint, spine, or entheseal) AND at least 3 points of the following categories:

   a) Evidence of psoriasis: (Score for one of the following) i) Current psoriasis - 2 points (Psoriatic skin or scalp disease present today as judged by a dermatologist or rheumatologist) ii) Personal history of psoriasis - 1 point (A history of psoriasis that may be obtained from the subject, family physician, dermatologist, rheumatologist, or other qualified health care provider) iii) Family history of psoriasis - 1 point (A history of psoriasis in a first- or second-degree relative according to subject report) b) Psoriatic nail dystrophy - 1 point i) Typical psoriatic nail dystrophy, including onycholysis, pitting, and hyperkeratosis, observed on current physical examination c) A negative test for rheumatoid factor - 1 point i) By any method except latex, but preferably by enzyme-linked immunosorbent assay (ELISA) or nephelometry, according to the local laboratory reference range d) Dactylitis: (Score for 1 of the following) i) Current dactylitis - 1 point (Swelling of an entire digit) ii) History of dactylitis - 1 point (A history of dactylitis recorded by a rheumatologist) e) Radiologic evidence of juxta-articular new bone formation - 1 point i) Ill-defined ossification near joint margins (but excluding osteophyte formation) on plain radiographs of the hand or foot.
5. Evidence of axial involvement (e.g., active inflammation, structural changes) that has been demonstrated by previous imaging techniques (e.g., radiography, MRI, CT), is considered indicative of axial disease by central reader assessment (2 readers and adjudicator).
6. Screening/baseline MRI demonstrates definite active inflammation on MRI of SIJ and/or spine (ASAS definition of positive MRI and ≥4 SIJ quadrants with BME and/or ≥4 vertebral units with BME (in the absence of degenerative disc disease at those discovertebral units with BME)) as determined by central readers.
7. Presence of chronic back pain in the 3 months prior to screening.
8. Active disease as defined by a BASDAI value of ≥4 and TBP score of ≥4 (on a 0-10 NRS scale) at screening and baseline.
9. History of an inadequate response to at least two different NSAIDs over a period of 4 weeks in total at the maximum recommended or tolerated doses, or intolerance/contraindication (e.g., allergic reaction, gastrointestinal symptoms or signs, severe arterial hypertension, etc.) for NSAIDs.
10. For all females of child-bearing potential: must not have a positive serum pregnancy test at the Screening Visit and must have a negative urine pregnancy test at Baseline prior to the first dose of study drug (local practices may require serum pregnancy testing at Baseline). Subjects with a borderline serum pregnancy test at Screening must have absence of clinical suspicion of pregnancy or other pathological causes of borderline results and a serum pregnancy test ≥3 days later to document continued lack of a positive result (unless prohibited by local requirements).

    1. Female subjects of childbearing potential must practice at least 1 protocol-specified method of birth control that is effective from Study Day 1 through at least 30 days after the last dose of study drug (local practices may require 2 methods of birth control). Female subjects of non-childbearing potential do not need to use birth control.
    2. Females must not be pregnant, breastfeeding, or considering becoming pregnant during the study and for approximately 30 days after the last dose of study drug. Females must commit to one of the following methods of highly effective birth control:

       * Combined (estrogen- and progestogen-containing) hormonal birth control (oral, intravaginal, transdermal, injectable) associated with inhibition of ovulation initiated at least 30 days prior to study baseline.
       * Progestogen-only hormonal birth control (oral, injectable, implantable) associated with inhibition of ovulation initiated at least 30 days prior to study baseline.
       * Bilateral tubal occlusion/ligation (can be via hysteroscopy, provided a hysterosalpingogram confirms success of the procedure) (For Japan: only bilateral tubal ligation).
       * Intrauterine device (IUD).
       * Intrauterine hormone-releasing system (IUS).
       * Vasectomized sexual partner (the partner has received medical confirmation of the surgical success of the vasectomy and is the sole sexual partner of the trial subject).
       * Practice true abstinence (unless not acceptable per local practices), defined as: refraining from heterosexual intercourse when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable).
11. If required per local practices, females of childbearing potential must commit to using 2 methods of contraception (either 2 highly effective methods or 1 highly effective method combined with 1 effective method). Effective methods of birth control are the following:

    * Progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action, initiated at least 30 days prior to baseline.
    * Male or female condom with or without spermicide.
    * Cap, diaphragm, or sponge with spermicide.
    * A combination of male condom with a cap, diaphragm, or sponge with spermicide (double barrier method).
    * In questionable cases of menopausal status, a blood sample with simultaneous levels of follicle stimulating hormone (FSH) above 40 U/l and estradiol below 30 pg/ml is confirmatory.
12. Subjects who are regularly taking NSAIDs or analgesics (including mild opioids) as part of their PsA therapy are required to be on a stable dose/dose regimen for at least 14 days prior to the baseline visit. If entering the study on concomitant tramadol, combination of acetaminophen/paracetamol and codeine or combination of acetaminophen/paracetamol and hydrocodone, and/or non-opioid analgesics, subject must be on stable dose(s) for at least 14 days prior to the baseline Visit. However, subject must not have used opioid analgesics (except for combination of acetaminophen/paracetamol and codeine or combination of acetaminophen/paracetamol and hydrocodone which are allowed) within 14 days prior to the BL Visit.
13. Subjects taking oral corticosteroids must be on an average daily and stable dose of ≤10mg/day prednisone or equivalent for at least 14 days prior to the baseline visit.
14. Subjects taking topical therapies (e.g., topical JAKi, salicylic acid preparations, corticosteroids, retinoids) are allowed, but must be on a stable dose at least 4 weeks prior to the BL visit.
15. Subjects entering the study on the following concomitant csDMARDs must be on a stable dose as indicated below for at least 28 days prior to the baseline Visit (in case of Leflunomide washout must be either 8 weeks or 4 weeks with a standard cholestyramine wash-out). A combination of up to 2 background csDMARDs is allowed EXCEPT the combination of methotrexate (MTX) and leflunomide.

    * MTX (≤ 25 mg/week); or
    * Sulfasalazine (SSZ) (≤ 3 g/day); or
    * Hydroxychloroquine (≤ 400 mg/day); or
    * Chloroquine (≤ 250 mg/day); or
    * Leflunomide (≤ 20 mg/day); or
    * Apremilast (≤ 60 mg/day)
16. Subjects must have been treated for ≥ 3 consecutive months prior to the study entry with DMARD therapy (including csDMARD and/or bDMARD) and/or for ≥4 weeks of NSAID therapy (if csDMARDs are not indicated for their axial disease, in accordance with local product label for PSA, or nr-axSpA/AS for the subset with purely axial disease), but continue to exhibit active SpA, or had to discontinue previous DMARD and/or NSAID treatment due to intolerability or toxicity, irrespective of treatment duration .

    1. Subjects recruited in Europe: Subjects must have previously been treated with one or more DMARD (csDMARD as defined in inclusion criterion 15, and/or bDMARD) and deemed to be inadequate responders and/or intolerant.
    2. Subjects recruited in the US: Subjects must be TNFi-IR. In this study, an IR to TNFi therapy will be defined as patients who discontinue TNFi due to lack of efficacy based on the investigators' assessment or intolerance (irrespective of treatment duration).
    3. Subjects recruited in Canada: Subjects must have previously been treated with one or more DMARD (csDMARD as defined in inclusion criterion 15, and/or bDMARD) and deemed to be inadequate responders and/or intolerant.

       * Up to 20 patients presenting with purely axial disease and current psoriasis (at the time of screening) may be included in the study. These patients may have had a past history of joint involvement, but do not currently require csDMARD therapy. In order to be deemed eligible, these patients must meet both the ASAS Classification Criteria for axSpA and the CASPAR criteria, as well as all other inclusion/exclusion criteria, including inadequate response to 2 NSAIDs (inclusion criterion #9 - all countries), bioDMARD (Canada), and TNFi (US). The ASAS Classification Criteria for axSpA are provided in Appendix A.
17. If subjects are currently taking bioDMARD therapy, they may be recruited after an appropriate wash-out period of bioDMARD prior to the screening MRI. Prior exposure to a bioDMARD is allowed for no more than 75 subjects, and prior exposure to a 2nd bioDMARD is allowed for no more than 30 subjects (one bioDMARD must include TNFi for US patients). Washout periods are as follows: 4 weeks for Etanercept, 8 weeks for Infliximab, 10 weeks for Adalimumab, Golimumab, Certolizumab and Ixekizumab, 12 weeks for Ustekinumab, Secukinumab, Guselkumab, and Abatacept, and 20 weeks for Risankizumab. However, subjects should not stop their previous successful biological therapy only to be included in this study. For patients intolerant to bioDMARD and not on such treatment a washout period may not be necessary.

Exclusion Criteria:

1. Active infection(s) requiring treatment with parenteral anti-infectives within 30 days, or oral anti-infectives within 14 days prior to the baseline Visit; Chronic recurring infection and/or active viral infection that based on the investigator's clinical assessment makes the subject an unsuitable candidate for the study.
2. Confirmed COVID-19: the baseline visit must be at least 14 days from onset of signs/symptoms or positive SARS-CoV-2 test; symptomatic subjects must have recovered, defined as resolution of fever without use of antipyretics and improvement in symptoms;
3. Suspected COVID-19: subjects with signs/symptoms suggestive of COVID-19, known exposure, or high-risk behavior should undergo molecular (e.g., PCR) testing to rule out SARS-CoV-2 infection or must be asymptomatic for 14 days from a potential exposure;
4. History of recurrent (more than one episode) herpes zoster or disseminated/multi-dermatomal (a single episode) herpes zoster or disseminated (a single episode) herpes simplex.
5. Primary or secondary immunodeficiency.
6. Current clinical signs and symptoms suggestive for tuberculosis.
7. Tuberculosis Interferon Gamma Release Assay (IGRA) serum test and abnormal chest x-ray (positive x-ray) suggestive of past or present tuberculosis (both at screening, may be accepted if performed within 180 days prior to screening). If the IGRA test is indeterminate the test should be repeated. If it remains indeterminate the patient should be considered positive. Patients with a positive Tuberculosis IGRA serum test but negative chest x-ray and without clinical symptoms suggestive for tuberculosis may participate in the study after initiation of standard prophylactic anti-tuberculous treatment according to the current local treatment guidelines. At least 2 weeks prophylactic treatment is considered necessary prior to study participation. Patients should not take rifampin concurrently with Upadacitinib.
8. Chronic infection with hepatitis B virus. At screening HBsAg and anti-HBc will be tested. Patients who are HBsAg positive will be excluded. In case of HBsAg negativity, but anti-HBc positivity, participation in the study is possible if HBV-DNA testing is negative and liver function tests are normal.
9. Chronic infection with hepatitis C (HCV) (HCV ribonucleic acid (RNA) detectable in any subject with anti-HCV antibody (HCV Ab), or Human Immunodeficiency Virus (HIV) infection confirmed by positive anti-HIV antibody test.
10. Female subjects who are breastfeeding, pregnant, or plan to become pregnant during the study or within 4 weeks following the last dose of study drug.
11. Subjects with chronic inflammatory articular disease (other than PsO or PsA or SpA), or systemic autoimmune diseases, e.g., systemic lupus erythematosus, Sjögren´s syndrome, RA, unequivocal chronic fatigue syndrome, or unequivocal fibromyalgia. Subjects with a diagnosis of Crohn's disease or ulcerative colitis are allowed as long as they have no active symptomatic disease within 4 weeks prior to BL.
12. Concomitant treatment with strong inductors or inhibitors of cytochrome P450 3A (e.g., Ketoconazole, Fluconazole, Rifampicin, Clarithromycin, St-John´s-wort).

    Strong CYP3A Inhibitors:
    * Boceprevir
    * Cobicistat
    * Clarithromycin
    * Conivaptan
    * Grapefruit (fruit or juice)
    * Indinavir
    * Itraconazole
    * Ketoconazole
    * Lopinavir/Ritonavir
    * Mibefradil
    * Nefazodone
    * Nelfinavir
    * Posaconazole
    * Ritonavir
    * Saquinavir
    * Telaprevir
    * Telithromycin
    * Troleandomycin
    * Voriconazole

    Strong CYP3A Inducers:
    * Carbamazepine
    * Phenytoin
    * Rifampin
    * Rifapentine
    * St. John's Wort

    Information regarding potential drug interactions with upadacitinib can be located in the upadacitinib Investigator's Brochure.
13. Prior treatment with upadacitinib or another JAK-inhibitor or TYK2-inhibitor.
14. History of hypersensitivity to any component of upadacitinib tablets.
15. Treatment with intravenous, intramuscular or intraarticular/periarticular, or intrarectal steroids within 4 weeks prior to baseline Visit; treatment with oral steroids in a dose of >10 mg prednisolone equivalent per day.
16. Subject must not have been treated with any investigational drug of chemical or biologic nature within a minimum of 30 days or five half-lives (whichever is longer) prior to the first dose of study drug or is currently enrolled in another interventional clinical study.
17. History of an infected joint prosthesis at any time, with the prosthesis still in situ.
18. Actual malignancies or history of malignancies with curative treatment within 5 years prior to screening, except successfully treated non-metastatic squamous cell or basal cell carcinoma of the cutis or carcinoma in situ of the cervix.
19. A subject with any condition possibly affecting oral drug absorption, e.g., gastrectomy, clinically significant diabetic gastroenteropathy, or certain types of bariatric surgery such as gastric bypass. Procedures such as gastric banding, that simply divides the stomach into separate chambers, are NOT exclusionary.
20. Significant trauma or surgery procedure within 4 weeks prior to baseline or any preplanned elective surgery during the study period.
21. Evidence of other severe uncontrolled gastrointestinal, hepatic (serum albumin <25 mg/l or Child-Pugh-Score >10), renal, pulmonary, cardiovascular, nervous or endocrine disorders.
22. Any history of prior cardiovascular event, including but not limited to cerebrovascular accident, myocardial infarction, coronary stenting, and aorto-coronary bypass surgery.
23. History of thrombosis and/or hematological disorder increasing the propensity to thrombosis.
24. Any subject who has been vaccinated with live or attenuated vaccines within the 4 weeks prior to the first dose of study medication or is to be vaccinated with these vaccines at any time during treatment or within 4 weeks after the last dose of study drug.

    * Examples of live vaccines include, but are not limited to, the following:

      1. Monovalent live influenza A (H1N1) (intranasal);
      2. Seasonal trivalent live influenza (intranasal);
      3. Zostavax (herpes zoster, live attenuated);
      4. Rotavirus;
      5. Varicella (chicken pox);
      6. Measles-mumps-rubella or measles-mumps-rubella-varicella;
      7. Oral polio vaccine;
      8. Smallpox;
      9. Yellow fever;
      10. Bacille Calmette-Guérin;
      11. Typhoid (oral).
    * Administration of inactivated (non-replicating) vaccines is permitted prior to or during the study according to local practice guidelines. Examples of common vaccines that are inactivated, toxoid or biosynthetic include, but are not limited to, injectable influenza vaccine, pneumococcal, Shingrix (zoster vaccine, recombinant, adjuvanted), pertussis (Tdap) vaccines, monkey pox vaccine and SARS-CoV-2 (inactivated, mRNA, RNA). Whenever possible, subjects should not have received a COVID-19 vaccination in the 7 days prior to randomization or plan to receive a COVID-19 vaccination within the first 7 days after initiation of study drug.
25. Any of the following lab abnormalities detected at screening:

    1. Hemoglobin <8 g/dl;
    2. Absolute neutrophil count <1.0 x 109/L (<1000/mm3)
    3. Absolute lymphocyte count <0.50 x 109/L (<750/mm3)
    4. Platelet count <100 x 109/L (<100,000/mm3).
26. Patients with contraindications for the MRI including but not limited to claustrophobia, seizure disorders, presence of an implanted electronic device (e.g. heart pacemaker, insulin pump, etc.) or metal implants not known to be MRI safe and metal foreign bodies in the patient's body suspected to be ferromagnetic, tattoos performed with metal-containing paints or tattoos of large skin areas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the (SPARCC) MRI inflammation score (for SIJ and spine) at 12 weeks of therapy with upadacitinib vs placebo in the DMARD-IR (conventional and/or biologic) subgroup | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS-CRP) at Week 12 with upadacitinib vs placebo in the DMARD-IR (conventional and/or biologic) subgroup | 12 weeks
Change from Baseline in BASDAI at Week 12 with upadacitinib vs placebo in the DMARD-IR (conventional and/or biologic) subgroup | 12 weeks
Change from baseline in the (SPARCC) MRI inflammation score (for SIJ and spine) at 12 weeks of therapy with upadacitinib vs placebo in the overall population (NSAID-IR, c-DMARD-IR and and bio-DMARD-IR) | 12 weeks
Change from baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS-CRP) at Week 12 with upadacitinib vs placebo in the overall population (NSAID-IR, c-DMARD-IR and and bio-DMARD-IR) | 12 weeks
Change from Baseline in BASDAI at Week 12 with upadacitinib vs placebo in the overall population (NSAID-IR, c-DMARD-IR and and bio-DMARD-IR) | 12 weeks
Incidence of Adverse Events (AEs), AEs leading to withdrawal from study drug, and serious AEs (SAEs). | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Walter Maksymowych, Dr., Principal Investigator — CARE ARTHRITIS LTD.
Locations (4):
- United States (2):
  - Oregon Health and Science University, Portland, Oregon
  - DM Clinical Research, Tomball, Texas
- Canada (2):
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - Groupe de Recherche en Maladies Osseuses (G.R.M.O.) Inc., Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided